CLINICAL TRIAL: NCT00966849
Title: The Scientific Evaluation of a Cash Transfer Pilot Project to Support Orphans and Vulnerable Children (OVC) in Manicaland, Zimbabwe
Brief Title: Manicaland Cash Transfer Trial for Children in Zimbabwe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Biomedical Research and Training Institute (Other); Catholic Relief Services (Other); UNICEF (Other); Wellcome Trust (Other); World Bank (Other)
Responsible Party: Principal Investigator, Simon Gregson, Professor, Imperial College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: inh051
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Vaccination; Education; Birth Registration; Financial Support
Keywords: Randomized Controlled Trial; Financial Support; Poverty; Child, Orphaned; HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conditional Cash Transfer (Experimental): Vulnerable households in this arm will receive conditional cash transfers. A standard agricultural package (e.g. seeds, fertiliser etc) will be made available. Parenting skills classes will also be made available. Standard social services will continue in the area.
  Interventions: Other: Conditional Cash Transfer; Other: Standard Agricultural Package; Other: Parenting Skills Classes
- Unconditional Cash Transfer (Experimental): Vulnerable households in this arm will receive unconditional cash transfers. A standard agricultural package (e.g. seeds, fertiliser etc) will be made available. Parenting skills classes will also be made available. Standard social services will continue in the area.
  Interventions: Other: Unconditional Cash Transfers; Other: Standard Agricultural Package; Other: Parenting Skills Classes
- Control (Other): Vulnerable households in this arm will not receive cash transfers. A standard agricultural package (e.g. seeds, fertiliser etc) will be made available. Parenting skills classes will also be made available. Standard social services will continue in the area.
  Interventions: Other: Standard Agricultural Package; Other: Parenting Skills Classes

INTERVENTIONS:
Other: Conditional Cash Transfer — Households will receive bimonthly payments of US$18 plus US$4 per child under 18 years living in the house up to a maximum of 3 children i.e. transfers will vary from $22 to $30. Households will only be given the cash if they comply with the following conditions:
  * An application for a birth certificate must be made for all children under 18 years in the household who do not already have a birth certificate, including all newborn children within 3 months of birth.
  * All children under 5 years in the household must be up-to-date with vaccinations.
  * All children under 5 years must attend a growth monitoring clinic twice per year.
  * All children 6-17 years in the household attended school at least 90% of days in the last month.
  * At least one adult from each household attended at least 2 of the 3 most recent parenting skills classes.
  Arms: Conditional Cash Transfer
Other: Unconditional Cash Transfers — Households will receive bimonthly payments of US$18 plus US$4 per child under 18 years living in the house up to a maximum of 3 children i.e. transfers will vary from $22 to $30. Households will not be required to comply with conditions in order to receive the cash.
  Arms: Unconditional Cash Transfer
Other: Standard Agricultural Package — A standard agricultural package (e.g. seeds, fertiliser etc.) will be distributed in all study arms including the control arm as a gesture of goodwill to all those participating in the study.
Other: Parenting Skills Classes — 2-3 parenting skills classes will be held annually in each study cluster.

SUMMARY:
The purpose of this study is to determine whether cash transfers (conditional and unconditional) can improve health and social outcomes amongst children living in vulnerable households in Manicaland, eastern Zimbabwe. The study hypotheses are:

1. Cash transfers will increase the percentage of vulnerable children aged 0-4 years with a birth certificate.
2. Cash transfers will increase the percentage of vulnerable children aged 0-4 years with up-to-date vaccinations.
3. Cash transfers will increase the percentage of vulnerable children aged 6-12 years attending primary school at least 80% of days per month.

DETAILED DESCRIPTION:
Cash transfer programmes provide cash to families caring for orphans and vulnerable children (OVC). Conditional cash transfer programmes require families to comply with conditions relating to child health, education and general social welfare in order to receive the cash.

We plan to evaluate conditional and unconditional cash transfer programmes in Manicaland, eastern Zimbabwe - a predominantly rural area with high HIV prevalence. We will employ a cluster randomised controlled trial design. Ten existing study sites that represent four socio-economic strata - subsistence farming areas, roadside trading settlements, large-scale agricultural estates (tea estates and forestry estates) and small towns - have been identified as part of a separate, ongoing cohort study. Each site has been divided into 3 smaller, socio-economically homogenous clusters providing a total of 30 clusters that will form ten matched triplets. One site from each matched triplet will then be randomly assigned to one of three study arms - conditional cash transfer arm, unconditional cash transfer arm, and standard social services arm.

Data on the primary endpoints will be collected using a rapid, baseline census of all households in the study clusters. This will take approximately 3 months to complete. The cash transfer programmes will commence, in the appropriate intervention arms, shortly after completion of baseline data collection. A similar follow-up census will take place two years after initiation of the intervention.

The cash transfer interventions will be delivered by a local NGO called Diocese of Mutare Community Care Programme (DOMCCP), who work in partnership with Catholic Relief Services Zimbabwe. The baseline and follow-up censuses will be managed and conducted by the Biomedical Research and Training Institute Zimbabwe (BRTI) and Imperial College London. Data will also be collected from children in a sample of households from each of the study clusters as part of the ongoing Manicaland Cohort Study, which is a parallel study conducted by BRTI and Imperial College London. This data will also be used to evaluate the cash transfer programmes.

ELIGIBILITY:
Inclusion Criteria:

A household will be defined as vulnerable and thereby eligible for inclusion in the programme if there are children <18 years resident in the household at baseline AND

* household is in the poorest quintile of households (20%) at baseline OR
* household contains one or more orphans at baseline OR
* the household head is under 18 years of age at baseline OR
* household contains a chronically ill member OR
* household contains a disabled member

A household will be defined as individuals that live within the same homestead and eat from the same pot.

Exclusion Criteria:

Households already receiving cash transfers for orphans or vulnerable children (OVC) will not be eligible to enroll in the pilot programme.

During the trial, households that do not qualify at baseline but whose conditions later change such that they become eligible to participate in the pilot will not be able to enroll.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4043 (Actual)
Dates: Start 2009-08; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Robertson, MSc, Principal Investigator — Imperial College London; Simon Gregson, DPhil, Principal Investigator — Imperial College London; Constance Nyamukapa, PhD, Principal Investigator — Imperial College London; Shungu Munyati, MSc, Principal Investigator — Biomedical Research and Training Institute; Phyllis Mushati, MSc, Principal Investigator — Biomedical Research and Training Institute
Locations (1):
- Biomedical Research and Training Institute, Harare, Zimbabwe

REFERENCES:
- [Background] Robertson L, Mushati P, Skovdal M, Eaton JW, Makoni JC, Crea T, Mavise G, Dumba L, Schumacher C, Sherr L, Nyamukapa C, Gregson S. Involving Communities in the Targeting of Cash Transfer Programs for Vulnerable Children: Opportunities and Challenges. World Dev. 2014 Feb;54(100):325-337. doi: 10.1016/j.worlddev.2013.09.002. PMID 24748713
- [Background] Robertson L, Mushati P, Eaton JW, Sherr L, Makoni JC, Skovdal M, Crea T, Mavise G, Dumba L, Schumacher C, Munyati S, Nyamukapa C, Gregson S. Household-based cash transfer targeting strategies in Zimbabwe: are we reaching the most vulnerable children? Soc Sci Med. 2012 Dec;75(12):2503-8. doi: 10.1016/j.socscimed.2012.09.031. Epub 2012 Oct 5. PMID 23103074
- [Result] Robertson L, Mushati P, Eaton JW, Dumba L, Mavise G, Makoni J, Schumacher C, Crea T, Monasch R, Sherr L, Garnett GP, Nyamukapa C, Gregson S. Effects of unconditional and conditional cash transfers on child health and development in Zimbabwe: a cluster-randomised trial. Lancet. 2013 Apr 13;381(9874):1283-92. doi: 10.1016/S0140-6736(12)62168-0. Epub 2013 Feb 27. PMID 23453283
- [Result] Crea TM, Reynolds AD, Sinha A, Eaton JW, Robertson LA, Mushati P, Dumba L, Mavise G, Makoni JC, Schumacher CM, Nyamukapa CA, Gregson S. Effects of cash transfers on Children's health and social protection in Sub-Saharan Africa: differences in outcomes based on orphan status and household assets. BMC Public Health. 2015 May 28;15:511. doi: 10.1186/s12889-015-1857-4. PMID 26017676
- [Result] Skovdal M, Robertson L, Mushati P, Dumba L, Sherr L, Nyamukapa C, Gregson S. Acceptability of conditions in a community-led cash transfer programme for orphaned and vulnerable children in Zimbabwe. Health Policy Plan. 2014 Oct;29(7):809-17. doi: 10.1093/heapol/czt060. Epub 2013 Sep 9. PMID 24019380
- [Result] Skovdal M, Mushati P, Robertson L, Munyati S, Sherr L, Nyamukapa C, Gregson S. Social acceptability and perceived impact of a community-led cash transfer programme in Zimbabwe. BMC Public Health. 2013 Apr 15;13:342. doi: 10.1186/1471-2458-13-342. PMID 23587136
- [Result] Fenton R, Nyamukapa C, Gregson S, Robertson L, Mushati P, Thomas R, Eaton JW. Wealth differentials in the impact of conditional and unconditional cash transfers on education: findings from a community-randomised controlled trial in Zimbabwe. Psychol Health Med. 2016 Dec;21(8):909-17. doi: 10.1080/13548506.2016.1140903. Epub 2016 Feb 22. PMID 26899880
- [Derived] Schaefer R, Thomas R, Robertson L, Eaton JW, Mushati P, Nyamukapa C, Hauck K, Gregson S. Spillover HIV prevention effects of a cash transfer trial in East Zimbabwe: evidence from a cluster-randomised trial and general-population survey. BMC Public Health. 2020 Oct 23;20(1):1599. doi: 10.1186/s12889-020-09667-5. PMID 33097016

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrolment number (4043) represents the total number of Households enrolled in the study
Units Other Than Participants: Households
Groups:
- Conditional Cash Transfer: Vulnerable households in this arm will receive conditional cash transfers. A standard agricultural package (e.g. seeds, fertiliser etc) will be made available. Parenting skills classes will also be made available. Standard social services will continue in the area.
  Conditional Cash Transfer: Households will receive bimonthly payments of US$18 plus US$4 per child under 18 years living in the house up to a maximum of 3 children i.e. transfers will vary from $22 to $30. Households will only be given the cash if they comply with the following conditions:
  * An application for a birth certificate must be made for all children under 18 years in the household who do not already have a birth certificate, including all newborn children within 3 months of birth.
  * All children under 5 years in the household must be up-to-date with vaccinations.
  * All children under 5 years must attend a growth monitoring clinic twice per year.
  * All children 6-17 years in the household attended school
Period: Overall Study
Arm/Group | Conditional Cash Transfer | Unconditional Cash Transfer | Control
Started | 3660; 1319 Households | 3976; 1525 Households | 3169; 1199 Households
Completed | 2119; 1248 Households | 2498; 1452 Households | 1876; 1118 Households
Not Completed | 1541; 71 Households | 1478; 73 Households | 1293; 81 Households

BASELINE CHARACTERISTICS:
Groups:
- Conditional Cash Transfer: Conditional Cash Transfer: Households will receive bimonthly payments of US$18 plus US$4 per child under 18 years living in the house up to a maximum of 3 children i.e. transfers will vary from $22 to $30. Households will only be given the cash if they comply with the following conditions:
  * An application for a birth certificate must be made for all children <18 years in the household who do not already have a birth certificate, including all newborn children within 3 months of birth.
  * All children <5 yrs in the household must be up-to-date with vaccinations
  * All children <5 yrs must attend a growth monitoring clinic twice per yr
  * All children 6-17 yrs in the household attended school at least 90% of days in the last month
  * At least one adult from each household attended at least 2/3 most recent parenting skills classes
  Other procedures will be the same as in the unconditional cash transfer arm.
- Total: Total of all reporting groups
Arm/Group | Conditional Cash Transfer | Unconditional Cash Transfer | Control | Total
Number analyzed (Participants) | 3660 | 3976 | 3169 | 10805
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3660 | 3976 | 3169 | 10805
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data on sex are only available for the age-groups to which the primary outcomes and conditions applied - i.e. 0-4 year-olds for birth registration and vaccinations; and 6-17 year-olds for school attendance.
  Participants
    number analyzed (Participants) | 2397 | 2661 | 2135 | 7193
    Female | 1179 | 1332 | 1064 | 3575
    Male | 1218 | 1329 | 1071 | 3618

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Children Under 5 Years in Vulnerable Households That Have a Birth Certificate
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Conditional Cash Transfer | Unconditional Cash Transfer | Control
Number analyzed (Participants) | 417 | 528 | 366
Participants | 252 | 255 | 163

2. Primary Outcome: Proportion of Children Under 5 Years in Vulnerable Households That Have Up-to-date Vaccinations
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Conditional Cash Transfer | Unconditional Cash Transfer | Control
Number analyzed (Participants) | 417 | 517 | 360
Participants | 317 | 393 | 253

3. Primary Outcome: Proportion of Children Aged 6-12 Years That Attended Primary School 80% of Days in the Last Month
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Conditional Cash Transfer | Unconditional Cash Transfer | Control
Number analyzed (Participants) | 889 | 1046 | 785
Participants | 772 | 895 | 608

4. Secondary Outcome: Proportion of Children Aged 13-17 Years That Attended Secondary School 80% of Days in the Last Month
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Conditional Cash Transfer | Unconditional Cash Transfer | Control
Number analyzed (Participants) | 811 | 922 | 722
Participants | 735 | 812 | 570

ADVERSE EVENTS:
Groups:
- Conditional Cash Transfer: Conditional Cash Transfer: Households will receive bimonthly payments of US$18 plus US$4 per child under 18 years living in the house up to a maximum of 3 children i.e. transfers will vary from $22 to $30. Households will only be given the cash if they comply with the following conditions:
  * An application for a birth certificate must be made for all children under 18 years in the household who do not already have a birth certificate, including all newborn children within 3 months of birth.
  * All children under 5 years in the household must be up-to-date with vaccinations.
  * All children under 5 years must attend a growth monitoring clinic twice per year.
  * All children 6-17 years in the household attended school at least 90% of days in the last month.
  * At least one adult from each household attended at least 2 of the 3 most recent parenting skills classes.
  Other procedures will be as described for the unconditional cash transfer arm.
Arm/Group | Conditional Cash Transfer | Unconditional Cash Transfer | Control
Serious Adverse Events (participants affected / at risk) | 0/3660 | 0/3976 | 0/3169
Other Adverse Events (participants affected / at risk) | 0/3660 | 0/3976 | 0/3169

LIMITATIONS AND CAVEATS:
The study was done shortly after a period of economic crisis in Zimbabwe which may limit this generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes